CLINICAL TRIAL: NCT04501614
Title: A Pivotal Phase 1/2, Single-Arm, Open-label Study to Evaluate the Safety and Efficacy of Ponatinib With Chemotherapy in Pediatric Patients With Philadelphia Chromosome-Positive (Ph+) Acute Lymphoblastic Leukemia (ALL) Who Have Relapsed or Are Resistant or Intolerant to a Prior Tyrosine Kinase Inhibitor-Containing Therapy, or Who Have the T315I Mutation
Brief Title: A Study of Ponatinib With Chemotherapy in Children, Teenagers, and Adults With Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase 1 enrollment was terminated due to dose-limiting toxicities, thus the study was terminated by Sponsor.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ponatinib-1501; 2019-002549-39 (EudraCT Number); U1111-1225-0394 (Other: WHO)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia (Ph+ALL); Ph+ Mixed Phenotype Acute Leukemia (MPAL); Philadelphia Chromosome-Like ALL (Ph-like ALL)
Keywords: Drug Therapy
MeSH Terms: interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ponatinib (Experimental): Ponatinib tablets, based on weight, in combination with chemotherapy backbone, orally, once daily in both reinduction block and consolidation block (35 days each including 29 days of treatment followed by rest period from chemotherapy for a minimum of 6 days consisting of daily ponatinib only) in Phase 1 to determine RP2D. In Phase 2 participants will receive ponatinib at RP2D in combination with chemotherapy backbone.
  Interventions: Drug: Ponatinib; Drug: Chemotherapy Agents

INTERVENTIONS:
Drug: Ponatinib — Ponatinib tablets.
Drug: Chemotherapy Agents — Chemotherapy agents for reinduction include vincristine, dexamethasone, polyethylene glycol (PEG)-asparaginase (Erwinia asparaginase when PEG-asparaginase is not available), daunorubicin. Agents for intrathecal (IT) chemotherapy, central nervous system (CNS)-1/2: IT methotrexate chemotherapy, or CNS-3: triple intrathecal (ITT) methotrexate, hydrocortisone, cytarabine. Chemotherapy agents for consolidation include dexamethasone, vincristine, methotrexate, PEG-asparaginase (Erwinia asparaginase when PEG-asparaginase is not available), cyclophosphamide, etoposide, CNS-1/2: IT methotrexate chemotherapy, CNS-3: ITT chemotherapy methotrexate, hydrocortisone, cytarabine. The doses for chemotherapy agents for reinduction will be given as per standard of care.

SUMMARY:
This study is about an anticancer drug called ponatinib which is a tyrosine kinase inhibitor given with chemotherapy to children, teenagers, and young adults up to 21 years of age with Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia who have relapsed or are resistant to other treatment.

The main aims of this study are to confirm the highest dose of ponatinib tablets and minitablet capsules that can be given to participants with acceptable side effects, and to evaluate if participant's leukemia achieves remission.

Participants will take ponatinib tablets with chemotherapy. For participants who cannot swallow tablets or who are receiving less than a 10 milligrams (mg) dose, a capsule with small ponatinib minitablets inside will be provided. Participants will take ponatinib for 10 weeks in combination with chemotherapy (reinduction and consolidation blocks) and will be followed up for at least 3 years.

DETAILED DESCRIPTION:
The drug being tested in this study is called ponatinib. Ponatinib is being tested to treat pediatric population who have Philadelphia chromosome-positive (Ph+) acute lymphoblastic leukemia (ALL), Ph+ mixed phenotype acute leukemia (Ph+ MPAL), or Philadelphia chromosome-like ALL who have relapsed or are resistant or intolerant to a prior tyrosine kinase inhibitor (TKI)-containing therapy, or who have the T315I mutation.

The study will enroll approximately 68 participants. Participants will be assigned to a treatment group either in phase 1 or phase 2. Participants unable to swallow the ponatinib tablets or who are receiving less than a 10 mg dose will receive the age-appropriate formulation, capsule with ponatinib minitablets inside:

• Ponatinib + Chemotherapy

All participants will be asked to take ponatinib once daily. In phase 1 ponatinib will be administered in combination with a chemotherapy backbone to determine the recommended phase 2 dose (RP2D) of ponatinib. In both phase 1 and phase 2, treatment consists of two 35-day blocks of therapy (reinduction block and consolidation block). Each block will include 29 days of treatment of daily ponatinib and a chemotherapy backbone regimen followed by a rest period from chemotherapy for a minimum of 6 days consisting of daily ponatinib only.

This is a multi-center trial and will be conducted worldwide. The overall time to participate in this study is 6.5 years. Participants will make multiple visits to the clinic, and may be contacted by telephone in at least 36 months of follow-up after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a diagnosis of Ph+ ALL, Philadelphia chromosome-positive plus mixed phenotype acute leukemia (Ph+ MPAL), or Ph-like ALL with:

   a) Involvement of BM with ALL, including one of the following: i. M2 BM (5%-24% lymphoblasts): by morphology with confirmatory testing consisting of at least one of the following: flow cytometry lymphoblasts ≥5%, or BCR-ABL1 fluorescence in situ hybridization, or ≥10-2 leukemic clone identified by immunoglobulin heavy chain-T-cell receptor polymerase chain reaction, OR ii. M3 BM (≥25% lymphoblasts): by morphology, OR iii. Participants with combined BM (as defined above) and extramedullary disease.

   b) Evidence of Ph+ ALL, MPAL, or Ph-like ALL: i. Definite evidence of BCR-ABL1 fusion (Ph) for Ph+ ALL and MPAL, OR ii. Definite evidence of Ph-like ALL with targetable kinase-activating lesions involving any of the following kinase genes: ABL1, ABL2, CSF1R, and PDGFRB.

   Ph-like ALL diagnosis requires the identification of specified targetable kinase-activating lesions preferably by ribonucleic acid (RNA) sequencing or by alternative accredited method used by the site.

   c) Disease status: (i) For non-US sites: participants who have relapsed (post 0 or 1 HSCT) or are resistant or intolerant to at least one prior therapy that contained a BCR-ABL-targeted tyrosine kinase inhibitor (TKI), or for US sites: participants who have relapsed (post 0 or 1 HSCT) or are resistant or intolerant to at least one prior therapy that contained a second-generation BCR-ABL1-targeted TKI (i.e, dasatinib, nilotinib, and bosutinib); OR (ii) Have a BCR-ABL1 T315I mutation irrespective of relapse, resistance/intolerance, or transplant status and irrespective of any prior TKI use.

   Notes:

   A participant will be defined as intolerant if they had a Grade ≥3 nonhematologic toxicity or a Grade 4 hematologic toxicity considered related to the last TKI and lasting for >2 weeks, and led to discontinuation of therapy.
2. Weight: Participants must be weighing at least 5 kg at the time of enrollment.
3. Performance Status: Karnofsky performance status ≥50% for participants ≥16 years of age or Lansky Play Scale ≥50% for participants <16 years of age.
4. Have recovered to less than Grade 2 National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) Version 5.0, or to baseline, from any nonhematologic toxicities (except alopecia) due to previous therapy.
5. Participants must meet the following criteria related to prior therapies:

   * Cytoreduction with hydroxyurea: Hydroxyurea can be initiated and continued for up to 24 hours before the start of protocol therapy.
   * Participants who relapsed while receiving cytotoxic therapy: At least 14 days must have passed since the completion of the last dose of chemotherapy before the first dose of ponatinib can be given except for the following: intrathecal (IT) chemotherapy and/or maintenance therapy such as vincristine, mercaptopurine, methotrexate, or glucocorticoids. There is no waiting period for those relapsing on maintenance-like therapy.
   * HSCT: Participants who have experienced relapse after a HSCT are eligible, provided they have no evidence of acute or chronic graft-versus-host disease (GVHD), are not receiving GVHD prophylaxis or treatment, and are at least 90 days posttransplant at the time of enrollment.
   * Hematopoietic growth factors: Before the first dose of ponatinib, at least 7 days must have passed since completion of therapy with granulocyte colony-stimulating factor or other growth factors, and at least 14 days must have passed since completion of therapy with pegfilgrastim.
   * Biologics and targeted therapies: Before the first dose of ponatinib, at least 7 days must have passed since the last dose of a biologic agent. For agents that have known AEs occurring beyond 7 days after administration, this period must be extended beyond the time during which AEs are known to occur. The duration of this interval must be discussed with the sponsor's medical monitor/designee.
   * Monoclonal antibodies: After the last dose of monoclonal antibody, at least 3 half-lives of the administered antibody must have passed before the first dose of ponatinib.
   * Immunotherapy: Before the first dose of ponatinib, at least 30 days must have passed after the completion of any type of immunotherapy (eg, tumor vaccines, chimeric antigen receptor T-cell [CAR-T-cell]).
   * Immunosuppressive therapy: Before the first dose of ponatinib, at least 14 days must have passed after the completion of immunosuppressive therapy (including regimens following stem cell transplant).
   * Radiotherapy: No washout period is necessary for radiation given to any extramedullary site other than central nervous system (CNS); ≥90 days must have passed if participant received prior total body irradiation or craniospinal or cranial radiotherapy.
   * Anthracyclines: Participants must have had a lifetime exposure of <400 milligrams per square meter (mg/m^2) of doxorubicin equivalents of anthracyclines.
6. a) Adequate renal function defined as: Estimated glomerular filtration rate (eGFR) using the Schwartz formula, OR radioisotope glomerular filtration rate (GFR)≥70 mL/min/1.73 m^2, OR a normal serum creatinine based on age and sex.

   b) Adequate liver function defined as: Direct bilirubin ≤1.5 times the upper limit of normal (ULN) for age AND ALT ≤5 times the ULN for age.
7. No clinical, radiological or laboratory evidence of pancreatitis, including:

   1. Serum lipase must be <2 times the ULN, AND
   2. Serum amylase must be <2 times the ULN.
8. Adequate cardiac function defined as shortening fraction ≥27% by echocardiogram (ECHO) OR left ventricular ejection fraction of ≥50% by ECHO or multigated acquisition scan (MUGA).
9. Normal QT interval with Fridericia correction method (QTcF) on screening electrocardiogram (ECG), defined as QTcF of ≤450 milliseconds (ms).

Exclusion Criteria:

1. A history or current diagnosis of Burkitt leukemia/lymphoma or mature B-cell leukemia.
2. A history or current diagnosis of chronic myeloid leukemia (CML).
3. Diagnosis of ALL, MPAL, or Ph-like ALL with targetable kinase-activating lesions after treatment with cytotoxic therapy for another cancer.
4. Diagnosis of another concurrent primary malignancy.
5. Clinically significant cardiovascular disease, including but not limited to:

   1. Any history of myocardial infarction (MI) or unstable angina.
   2. History of or presence of heart block, and/or clinically significant ventricular or atrial arrhythmias.
   3. Uncontrolled hypertension, defined as persistent elevation of systolic and/or diastolic blood pressures to ≥95th percentile based on age, sex, and height percentiles despite appropriate antihypertensive management.
6. Current systemic use of drug(s) that are known to have a risk of causing prolonged corrected QT interval (QTc) or torsades de pointes unless drug(s) can be changed to acceptable alternatives (ie, an alternate class of agents that do not affect the cardiac conduction system) or the participants can safely discontinue the drug(s).
7. Uncontrolled hypertriglyceridemia (triglycerides ≥450 milligrams per deciliter (mg/dL)).
8. Current systemic use of any medications or herbal supplements that are known to be strong inhibitors or strong inducers of cytochrome P450 3A (CYP3A) within 7 days before the first dose of study drug.
9. Previous treatment with ponatinib.
10. Planned non-protocol chemotherapy, radiation therapy, another investigational agent, or immunotherapy while participant is on study treatment.
11. Known gastrointestinal disease or gastrointestinal procedure that could interfere with the oral absorption of ponatinib.
12. Participants with deoxyribonucleic acid (DNA) fragility syndromes, such as Fanconi anemia and Bloom syndrome.
13. Participants with Down syndrome.
14. Participants with uncontrolled systemic infection, or known laboratory and/or clinical evidence of active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
15. Participants with pre-existing significant CNS pathology, including history of severe brain injury, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination/movement disorder, or autoimmune disease with CNS involvement, are not eligible.
16. Participants with a history of cerebrovascular ischemia/hemorrhage with residual deficits are not eligible. (Participants with a history of cerebrovascular ischemia/hemorrhage remain eligible provided all neurologic deficits and causative factor(s) have resolved).
17. Uncontrolled seizure disorder. (Participants with seizure disorders that do not require antiepileptic drugs or are well controlled with stable doses of antiepileptic drugs are eligible).
18. History of severe coagulopathy or cardiovascular or peripheral vascular events.
19. Treatment with live attenuated vaccinations within 30 days prior to initiation of study treatment regimen.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (64):
- United States (13):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Childrens Hospital San Diego - PIN, San Diego, California
  - UCSF Medical Comprehensive Cancer, San Francisco, California
  - Alfred I Dupont Hospital For Children, Wilmington, Delaware
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Riley Hospital For Children, Indianapolis, Indiana
  - Children's Mercy Hospital and Clinica, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center - PIN, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Childrens Medical Center Research Institute at UT Southwestern, Dallas, Texas
- Argentina (2):
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
- Australia (3):
  - Queensland Childrens Hospital, South Brisbane, Queensland
  - Royal Children's Hospital Melbourne - PIN, Parkville, Victoria
  - Perth Childrens Hospital, Nedlands, Western Australia
- Brazil (7):
  - Rua Ramiro Barcelos, 2350, Curitiba, Paraná
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande Du Sul
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande Du Sul
  - Fundacao Pio XII Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP, Ribeirão Preto
  - Graacc Grupo de Apoio Ao Adolescente E A Crianca Com Cancer, São Paulo
  - Hospital Santa Marcelina, São Paulo
- China (11):
  - West China Second University Hospital, Sichuan Univesity, Chengdu
  - Children's Hospital of Chongqing Medical University, Chongqing
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second Hospital of Anhui Medical University, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - Children's Hospital of Shanghai, Shanghai
  - Shanghai Childrens Medical Center, Shanghai
  - Children's Hospital of Soochow University, Suzhou
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice v Motole, Prague
- France (4):
  - Hopital Sud, Rennes, Ille-et-Vilaine
  - Assistance Publique Hopitaux de Marseille, Marseille
  - Hopital Robert Debre, Paris
  - Hopital Des Enfants, Toulouse
- Italy (4):
  - IRCCS Ospedale Pediatrico Bambino Gesu - INCIPIT - PIN, Rome, Lazio
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genoa, Liguria
  - Fndazione MBBM (MONZA E BRIANZA PER IL BAMBINO E LA SUA MAMMA) - c/o Centro Maria Letizia Verga, Monza, Lombardy
  - Ospedale Infantile Regina Margherita - INCIPIT - PIN, Turin, Piedmont
- Mexico (3):
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Nuevo Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara
  - Instituto Nacional de Pediatria, Mexico City
- Princess Maxima Center for Pediatric Oncology - PIN, Utrecht, Netherlands
- Poland (2):
  - Uniwersytecki Szpital Dzieciecy, Krakow
  - SPSK Nr 1 im. Prof.Stanislawa Szyszko Slaskiego Uniwersytetu Medycznego, Zabrze
- Portugal (2):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon, Lisbon District
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center - PPDS, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (3):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Infantil Universitario Nino Jesus - PIN, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- United Kingdom (3):
  - Royal Marsden Hospital - Surrey, Surrey Quays, Sutton
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Hospital for Children (Glasgow) - PPDS - PIN, Glasgow

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be reidentified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f929169296beb001e63bf5d

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of Philadelphia Chromosome-Positive (Ph+) Acute Lymphoblastic Leukemia (ALL) took part in the study at various investigative sites globally from 24 February 2021 to 19 July 2024.
Pre-assignment Details: Participants were enrolled in Phase 1 and received ponatinib per protocol specifications (presented per dose regimen here). Due to the observation of multiple dose-limiting toxicities (DLTs) in Phase 1, study enrollment was terminated per protocol and no recommended phase 2 dose (RP2D) could be determined. The Sponsor terminated the study following a 6-month follow-up and no participants were enrolled in Phase 2 of the study, thus, no Phase 2 results are presented here as it was not conducted.
Groups:
- Ponatinib 30 mg Adult-Equivalent: Participants received weight-based dose of ponatinib tablets 30 milligrams (mg) adult-equivalent, orally, once daily in combination with chemotherapy backbone per standard regimen at the investigator's discretion in both reinduction block and consolidation block (35 days each including 29 days of treatment in combination with chemotherapy followed by a minimum 6-day rest period from chemotherapy with daily ponatinib only) up to Day 70 (end of consolidation) followed by optional ponatinib continuation in Phase 1.
- Ponatinib 15 mg Adult-Equivalent: Participants received weight-based dose of ponatinib tablets 15 mg adult-equivalent, orally, once daily in combination with chemotherapy backbone per standard regimen at the investigator's discretion in both reinduction block and consolidation block (35 days each including 29 days of treatment in combination with chemotherapy followed by a minimum 6-day rest period from chemotherapy with daily ponatinib only) up to Day 70 (end of consolidation) followed by optional ponatinib continuation in Phase 1.
Period: Overall Study
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent
Started | 7 | 4
Completed | 0 | 0
Not Completed | 7 | 4
Not completed — Study Terminated by Sponsor | 6 | 3
Not completed — Withdrawal by Participant (Parent/Legal Guardian) | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received at least 1 dose of ponatinib.
Groups:
- Ponatinib 30 mg Adult-Equivalent: Participants received weight-based dose of ponatinib tablets 30 mg adult-equivalent, orally, once daily in combination with chemotherapy backbone per standard regimen at the investigator's discretion in both reinduction block and consolidation block (35 days each including 29 days of treatment in combination with chemotherapy followed by a minimum 6-day rest period from chemotherapy with daily ponatinib only) up to Day 70 (end of consolidation) followed by optional ponatinib continuation in Phase 1.
- Total: Total of all reporting groups
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (2.41) | 13.5 (3.70) | 12.6 (2.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D) of Ponatinib in Combination With Chemotherapy
Description: The RP2D is the maximum tolerated dose (MTD) or less.
Time Frame: Up to Day 35 in Phase 1
Population: The Safety Population included all participants who received at least 1 dose of ponatinib.
Measure: Number; unit: milligrams per square meter (mg/m^2)
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent
Number analyzed (Participants) | 7 | 4
milligrams per square meter (mg/m^2) | NA — Due to DLTs observed in both dose cohorts, study enrollment was terminated per protocol and participants were discontinued from study treatment per independent data monitoring committee (IDMC) advice followed by study termination by Sponsor. Thus, the RP2D could not be determined. | NA — Due to DLTs observed in both dose cohorts, study enrollment was terminated per protocol and participants were discontinued from study treatment per independent data monitoring committee (IDMC) advice followed by study termination by Sponsor. Thus, the RP2D could not be determined.

2. Primary Outcome: Phase 2: Percentage of Participants With Complete Remission (CR) at the End of the Reinduction Block
Description: CR was defined as no circulating blasts and less than (<)5 percent (%) blasts in the bone marrow (BM); normal maturation of all cellular components in the bone marrow; no extramedullary disease; absolute neutrophil count (ANC) greater than (>)1000 cells/microliter (μL) (or >1.0 × 10^9 cells/liter [L]); Platelets >100,000/μL (or >100 × 10^9 platelets/L).
Time Frame: Up to Day 35 in Phase 2
Population: The study enrollment was terminated per protocol due to DLTs observed in both dose cohorts in Phase 1 and the RP2D could not be determined leading to study termination by the Sponsor before Phase 2 could be initiated. No data was collected as no participants were enrolled in Phase 2.
Groups:
- Ponatinib RP2D: Participants were planned to receive weight-based dose of ponatinib tablets at the RP2D adult-equivalent, orally, once daily in combination with chemotherapy backbone per standard regimen at the investigator's discretion in both reinduction block and consolidation block (35 days each including 29 days of treatment in combination with chemotherapy followed by a minimum 6-day rest period from chemotherapy with daily ponatinib only) followed by optional ponatinib continuation with or without chemotherapy in Phase 2.
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 1: Number of Participants With CR at the End of Reinduction Block
Description: CR was defined as no circulating blasts and <5% blasts in the BM; normal maturation of all cellular components in the bone marrow; no extramedullary disease; ANC >1000 cells/μL (or >1.0 × 10^9 cells/L); Platelets >100,000/μL (or >100 × 10^9 platelets/L).
Time Frame: Day 35 in Phase 1
Population: The Safety Population included all participants who received at least 1 dose of ponatinib. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent
Number analyzed (Participants) | 6 | 3
Participants | 1 | 2

4. Secondary Outcome: Phase 2: Percentage of Ph+ ALL Participants Who Achieved CR at the End of Consolidation Block
Description: CR was defined as no circulating blasts and <5% blasts in the bone marrow; normal maturation of all cellular components in the bone marrow; no extramedullary disease; ANC >1000 cells/μL (or >1.0 × 10^9 cells/L); Platelets >100,000 platelets/μL (or >100 × 10^9 platelets/L).
Time Frame: Day 70 in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 2: Percentage of Ph+ ALL Participants With Negative Minimal Residual Disease (MRD) Among Those Who Achieved CR
Description: MRD negative rate is the percentage of participants who achieve MRD negative status by evaluation of bone marrow aspirate at <0.01% threshold.
Time Frame: Up to Day 70 (end of consolidation block) in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 2: Percentage of Participants Who Relapsed or Progressed Following Reinduction and Consolidation
Time Frame: Up to 3 years of follow-up in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 2: Event-free Survival (EFS)
Description: EFS was defined as time from date of enrollment until death due to any cause; refractory to treatment (defined as failure to achieve CR by end of the consolidation block) or relapse from CR. CR was defined as no circulating blasts and <5% blasts in the bone marrow; normal maturation of all cellular components in the bone marrow; no extramedullary disease; ANC >1000 cells/μL (or >1.0 × 10^9 cells/L); Platelets >100,000 platelets/μL (or >100 × 10^9 platelets/L).
Time Frame: Up to 3 years of follow-up in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as time from date of enrolment until death related to disease under study; disease progression (clinical deterioration associated with disease process, including evidence of increasing blasts in the bone marrow from baseline and/or evidence of new organ involvement) or relapse from CR. CR was defined as no circulating blasts and <5% blasts in the bone marrow; normal maturation of all cellular components in the bone marrow; no extramedullary disease; ANC >1000 cells/μL (or >1.0 × 10^9 cells/L); Platelets >100,000 platelets/μL (or >100 × 10^9 platelets/L).
Time Frame: Up to 3 years of follow-up in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as time from first dose of ponatinib until death due to any cause.
Time Frame: Up to 3 years of follow-up in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was defined as the interval between the first assessment at which the criteria for CR are met until the time at which relapse from CR occurs. CR was defined as no circulating blasts and <5% blasts in the bone marrow; normal maturation of all cellular components in the bone marrow; no extramedullary disease; ANC >1000 cells/μL (or >1.0 × 10^9 cells/L); Platelets >100,000 platelets/μL (or >100 × 10^9 platelets /L).
Time Frame: Up to 3 years of follow-up in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase 2: Percentage of Participants Who Underwent Hematopoietic Stem Cell Transplantation (HSCT)
Time Frame: Up to 3 years of follow-up in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase 1: Cmax: Maximum Observed Plasma Concentration for Ponatinib
Time Frame: Predose and at multiple timepoints post-dose up to 24 hours on Days 1 and 22 in Phase 1
Population: The Pharmacokinetic (PK) Analysis Population included all participants in the Phase 1 portion of the study who had sufficient ponatinib dosing data and concentration-time data to permit the calculation of ponatinib PK parameters. Number analyzed is the number of participants with data available for analysis for the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent
Number analyzed (Participants) | 7 | 4
nanograms/milliliter (ng/mL)
  Day 1 | 65.8 (29.5) | 24.9 (71.1)
  Day 22: number analyzed (Participants) | 1 | 2
  Day 22 | 183 (NA) — Geometric coefficient of variation (CV) was not estimable for a single participant. | 47.7 (92.8)

13. Secondary Outcome: Phase 1: Tmax: Time of First Occurrence of Cmax for Ponatinib
Time Frame: Predose and at multiple timepoints post-dose up to 24 hours on Days 1 and 22 in Phase 1
Population: The PK Analysis Population included all participants in the Phase 1 portion of the study who had sufficient ponatinib dosing data and concentration-time data to permit the calculation of ponatinib PK parameters. Number analyzed is the number of participants with data available for analysis for the specified timepoint.
Measure: Median (Full Range); unit: hours
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent
Number analyzed (Participants) | 7 | 4
hours
  Day 1 | 6.00 [2.0 to 7.5] | 3.99 [3.8 to 4.1]
  Day 22: number analyzed (Participants) | 1 | 2
  Day 22 | 4.08 [NA to NA] — Full range was not estimable for a single participant. | 3.92 [2.0 to 5.8]

14. Secondary Outcome: Phase 1: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Ponatinib
Time Frame: Predose and at multiple timepoints post-dose up to 24 hours on Days 1 and 22 in Phase 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter (h*ng/mL)
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent
Number analyzed (Participants) | 7 | 4
hours*nanograms/milliliter (h*ng/mL)
  Day 1 | 883 (22.8) | 264 (62.1)
  Day 22: number analyzed (Participants) | 1 | 2
  Day 22 | 2800 (NA) — Geometric CV was not estimable for a single participant. | 815 (83.2)

15. Secondary Outcome: Phase 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, Venous Thrombotic/Embolic Events (VTEs), and Adverse Events of Special Interest (AESIs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in clinical study participant, temporally associated with use of study intervention, whether or not occurrence was considered related to the study intervention including any unfavorable & unintended sign (e.g., clinically significant abnormal laboratory finding), symptom/disease. TEAE: any AE that occurs after administration of first dose of any study drug & through 30 days after last dose of any study drug. Serious TEAE:AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization/prolongation of existing hospitalization, resulted in persistent/significant disability or incapacity, was congenital anomaly/birth defect, was medically important event. AESI: Protocol-defined AEs resulting in compromise of organ function or other significant consequences. VTEs were identified as AESIs for ponatinib and included arterial, VTEs that meet criteria for serious TEAEs.
Time Frame: Up to 34.8 months in Phase 1
Population: The Safety Population included all participants who received at least 1 dose of ponatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent
Number analyzed (Participants) | 7 | 4
Participants
  TEAEs | 7 | 4
  Serious TEAEs | 5 | 2
  VTEs | 0 | 0
  AESIs | 0 | 0

16. Secondary Outcome: Phase 2: Number of Participants With TEAEs, Serious TEAEs, VTEs, and AESIs
Description: An AE is defined as any untoward medical occurrence in clinical study participant, temporally associated with use of study intervention, whether or not occurrence was considered related to the study intervention including any unfavorable & unintended sign (e.g., clinically significant abnormal laboratory finding), symptom/disease. TEAE: any AE that occurs after administration of first dose of any study drug & through 30 days after last dose of any study drug. Serious TEAE:AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization/prolongation of existing hospitalization, resulted in persistent/significant disability or incapacity, was congenital anomaly/birth defect, was medically important event. AESI: Protocol-defined AEs resulting in compromise of organ function or other significant consequences. VTEs were identified as AESIs for ponatinib and included arterial, VTEs that meet criteria for serious TEAEs.
Time Frame: Up to 30 days after last dose of ponatinib in Phase 2
Population: as for outcome 2
Arm/Group | Ponatinib RP2D
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 34.8 months in Phase 1
Description: The Safety Population included all participants who received at least 1 dose of ponatinib. The study was terminated following the Sponsor's decision attributed to DLTs observed in Phase 1. Hence, no participants were enrolled in Phase 2 of the study and no data for the same could be presented.
Arm/Group | Ponatinib 30 mg Adult-Equivalent | Ponatinib 15 mg Adult-Equivalent
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/7 | 2/4
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ponatinib 30 mg Adult-Equivalent (N=7) | Ponatinib 15 mg Adult-Equivalent (N=4)
Alanine aminotransferase increased (Investigations) | 2 | 1
Bilirubin conjugated increased (Investigations) | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ventricle dilatation (Nervous system disorders) | 1 | 0
Disseminated mucormycosis (Infections and infestations) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Seizure (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ponatinib 30 mg Adult-Equivalent (N=7) | Ponatinib 15 mg Adult-Equivalent (N=4)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Agitation (Psychiatric disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 4
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 4
Anal erythema (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Antithrombin III decreased (Investigations) | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 3
Asthenia (General disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bilirubin conjugated increased (Investigations) | 1 | 2
Blood albumin decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 4 | 1
Blood bilirubin unconjugated increased (Investigations) | 2 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood fibrinogen decreased (Investigations) | 4 | 1
Blood glucose increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Disseminated mucormycosis (Infections and infestations) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 3
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Eosinophil count decreased (Investigations) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Gallbladder oedema (Hepatobiliary disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 6 | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gingival erythema (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 5 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0
Monocyte count increased (Investigations) | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myringitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Neutrophil count decreased (Investigations) | 5 | 3
Neutrophil count increased (Investigations) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0
Oral infection (Infections and infestations) | 2 | 0
Pain (General disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Parotitis (Infections and infestations) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Platelet count decreased (Investigations) | 4 | 3
Platelet count increased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Protein total decreased (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 2
Swelling (General disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0
Ventricular hypertrophy (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1
White blood cell count decreased (Investigations) | 4 | 3
White blood cells urine positive (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT04501614/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04501614/SAP_001.pdf